CLINICAL TRIAL: NCT03307798
Title: Evaluate a Saw Bone Training Protocol in Using Tactile Sensation to Classify Bone Quality During Implant Surgery
Acronym: SBTP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201612189RIND
Record Dates: First submitted 2017-09-21; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-03

CONDITIONS: Surgery; Training Tactile Sensation; Diagnosis of Bone Quality
Keywords: dental implant,bone quality,tactile sensation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bone quality is one of the major factors influencing the dental implant survival rate. Bone quality is believed to have effects on initial implant stability and success of osseointegration. Different implant designs and surgical protocols were developed for improving the survival rate in different bone quality. Although bone quality can be partly diagnosed by radiographic images, lots of experienced surgeons also evaluate bone quality with tactile sensation when they drill the bone. However, variations in evaluation of bone density maybe exist among different surgeons. For less experienced dentists, it is difficult to diagnose bone quality with tactile sensation in the beginning. This purpose of this study is to evaluate a training protocol in using tactile sensation to classify bone quality during implant surgery. Saw bones of variant densities are used as training materials. The outcomes before and after training will be compared. The effect of training frequency before surgery will also be evaluated.

DETAILED DESCRIPTION:
Twenty-five dentists will be enrolled into the study. Tests will be performed using visual analog scale to score bone quality of test blocks.

ELIGIBILITY:
Inclusion Criteria:

* Certified dentist with implant surgery experience less than 10 implants.

Exclusion Criteria:

* Age exceed the limits
* Implant surgery experience more or equal to 10 implants

Ages: 26 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dentists in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Change on visual analog scale (VAS) score of each test block | 1st time point: test before training & test immediately after training; 2nd time point: 1 week after 1st time point (test after 1 wk); 3rd time point: 1 month after 2nd time point (test after 1month)
  Each VAS score performed on the specific test block will be compared between different time point.

CONTACTS AND LOCATIONS:
Overall Officials: Tong-Mei Wang Wang, DDS, MS, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Friberg B, Sennerby L, Meredith N, Lekholm U. A comparison between cutting torque and resonance frequency measurements of maxillary implants. A 20-month clinical study. Int J Oral Maxillofac Surg. 1999 Aug;28(4):297-303. PMID 10416900
- [Background] Johansson P, Strid KG. Assessment of bone quality from cutting resistance during implant surgery. Internatioanl Journal of Oral & Maxillofacial implants 9:279-288, 1994